CLINICAL TRIAL: NCT02713737
Title: Impact of High-flow Nasal Cannula Oxygen (HFNC) Versus Noninvasive Ventilation Associated With Sleep Quality on Atrial Fibrillation in Hypoxemic Patients After Coronary Surgery
Brief Title: The Correlation Between Sleep Quality and Atrial Fibrillation Undergoing High-flow Nasal Cannula Oxygen (HFNC)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Principal Investigator, Jian Zhao, associate professor, Henan Institute of Cardiovascular Epidemiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanICE; HenanICE201601 (Registry Identifier: HenanICE201601)
Record Dates: First submitted 2016-02-25; First posted 2016-03-21 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Hypoxemia
Keywords: hypoxemia; high-flow; atrial fibrillation; sleep
MeSH Terms: conditions — Hypoxia; Atrial Fibrillation | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HFNC group (Experimental): HFNC: Heated humidified high-flow nasal cannula.
  Interventions: Device: heated humidified high-flow nasal cannula
- NIV group (Active Comparator): NIV: Noninvasive ventilation.
  Interventions: Device: noninvasive ventilation

INTERVENTIONS:
Device: heated humidified high-flow nasal cannula — HFNC device (Airvo™, Fisher＆Paykel, Auckland, New Zealand) with a heated circuit (Fisher＆Paykel,900PT501) and nasal cannula(optiflow TM,Fisher＆Paykel). It has adjustable FiO2: 21%-100%, gas flow up to 60 L/min, to maintain arterial blood hemoglobin oxygen saturation ( SPO2) > 92%.
  Arms: HFNC group
Device: noninvasive ventilation — TBird VELA ventilator, CareFusion, USA. Pressure adjustments were to optimize patient comfort. Inspiratory pressure was raised every 5 mins until comfort was optimized. FiO2 was adjusted to maintain SPO2 > 92%.
  Other Names: noninvasive positive pressure ventilation
  Arms: NIV group

SUMMARY:
The investigators hypothesized that heated humidified high-flow nasal cannula oxygen(HFNC) along with high quality of sleep, in comparison with noninvasive positive pressure ventilation (NIV), could reduce the release of inflammatory marker C-reactive protein(CRP), which as independent predictor of atrial fibrillation（AF）, further lower the incidence of new-onset AF following coronary artery bypass grafting(CABG).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) has been reported to occur in up to 20-40% of patients undergoing coronary artery bypass grafting (CABG). Postoperative AF plays a major role in the determination of hemodynamic deterioration and can be associated with thromboembolic stroke. Aside from the risk factors of age, pain, cardiac dysfunction and hypokalemia, hypoxemia is also considered to be the major contributor to AF initiation and persistence. Aiming to the common postoperative complications, noninvasive positive pressure ventilation (NIV) provides an available modality to improve the oxygen and even obviate the reintubation.

However, some patients are contraindications for NIV, with Loss of consciousness, hemodynamic instability, and some are intolerance due to dryness, gastric distension, skin breakdown and noise, with complaints of insomnia and sleep disturbance. The aforementioned factors largely limits its use. Recently, the heated humidified high-flow nasal cannula (HFNC), free of psychic stress and physical discomfort, shows a favorable compliance and tolerance in treating the hypoxemic patients. As a result, in this comfortable setting we predict a high sleep quality in HFNC oxygen therapy. Evidence has suggested that sleep abnormalities trigger the cascaded release of C-reactive protein (CRP). As is well known that CRP is involved in atrial structural remodeling and asynchronous conduction, which attribute to the initiation and maintenance of AF.

Therefore, in this present study, the investigators first evaluate the sleep quality (architecture and duration) by the polysomnographic (PSG) monitoring after coronary surgery. Based on the sleep parameters, the investigators hypothesize that HFNC, along with high quality of sleep, in comparison with NIV, could reduce the release of C-reactive protein, which as independent predictor of atrial fibrillation (AF), further lower the incidence of new-onset AF following CABG.

ELIGIBILITY:
Inclusion criteria:

Hypoxemic respiratory failure

Exclusion criteria:

Cardiac or respiratory arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-04; Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of atrial fibrillation | 10 days
  from ICU admission to discharge

SECONDARY OUTCOMES:
PO2/FiO2(P/F) | 5 days
  from ICU admission to discharge
Lactate levels | 5 days
  from ICU admission to discharge
intubation time | 5 days
  from intubation in the operating room to discharge
transfusion requirement | 5 days
  from ICU admission to discharge
inotropic usage | 5 days
  from ICU admission to discharge
total sleep time | 48 hours
  The duration from 8 in the evening to 8 in the morning within the first 2 days after surgery.
rapid eye movement (REM) sleep (%) | 48 hours
  The duration from 8 in the evening to 8 in the morning within the first 2 days after surgery.
arousal index | 48 hours
  The duration from 8 in the evening to 8 in the morning within the first 2 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoyun Cheng, MD, Study Director — Henan Provincial People' Hospital
Locations (1):
- Henan Provincial People' Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meier-Ewert HK, Ridker PM, Rifai N, Regan MM, Price NJ, Dinges DF, Mullington JM. Effect of sleep loss on C-reactive protein, an inflammatory marker of cardiovascular risk. J Am Coll Cardiol. 2004 Feb 18;43(4):678-83. doi: 10.1016/j.jacc.2003.07.050. PMID 14975482
- [Background] Chanques G, Constantin JM, Sauter M, Jung B, Sebbane M, Verzilli D, Lefrant JY, Jaber S. Discomfort associated with underhumidified high-flow oxygen therapy in critically ill patients. Intensive Care Med. 2009 Jun;35(6):996-1003. doi: 10.1007/s00134-009-1456-x. Epub 2009 Mar 18. PMID 19294365
- [Background] Ucar HI, Tok M, Atalar E, Dogan OF, Oc M, Farsak B, Guvener M, Yilmaz M, Dogan R, Demircin M, Pasaoglu I. Predictive significance of plasma levels of interleukin-6 and high-sensitivity C-reactive protein in atrial fibrillation after coronary artery bypass surgery. Heart Surg Forum. 2007;10(2):E131-5. doi: 10.1532/HSF98.20061175. PMID 17597037
- [Background] Cuquemelle E, Pham T, Papon JF, Louis B, Danin PE, Brochard L. Heated and humidified high-flow oxygen therapy reduces discomfort during hypoxemic respiratory failure. Respir Care. 2012 Oct;57(10):1571-7. doi: 10.4187/respcare.01681. Epub 2012 Mar 12. PMID 22417569
- [Background] Elliott R, Rai T, McKinley S. Factors affecting sleep in the critically ill: an observational study. J Crit Care. 2014 Oct;29(5):859-63. doi: 10.1016/j.jcrc.2014.05.015. Epub 2014 May 29. PMID 24973105
- [Background] Stephan F, Barrucand B, Petit P, Rezaiguia-Delclaux S, Medard A, Delannoy B, Cosserant B, Flicoteaux G, Imbert A, Pilorge C, Berard L; BiPOP Study Group. High-Flow Nasal Oxygen vs Noninvasive Positive Airway Pressure in Hypoxemic Patients After Cardiothoracic Surgery: A Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2331-9. doi: 10.1001/jama.2015.5213. PMID 25980660
- [Result] Liu T, Li G, Li L, Korantzopoulos P. Association between C-reactive protein and recurrence of atrial fibrillation after successful electrical cardioversion: a meta-analysis. J Am Coll Cardiol. 2007 Apr 17;49(15):1642-1648. doi: 10.1016/j.jacc.2006.12.042. Epub 2007 Apr 2. PMID 17433956